CLINICAL TRIAL: NCT05804175
Title: Advanced Prediction of Respiratory Depression Episode With the Linshom Continuous Predictive Respiratory Sensor
Status: Recruiting | Type: Observational
Sponsor: Linshom Medical, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022H0375; R44HL164222 (NIH)
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Post Surgical Respiratory Failure; Respiratory Complication
Keywords: respiratory; monitoring; pulse oximetry; capnography; Linshom
MeSH Terms: interventions — Oximetry; Capnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Post surgical (non-cardiac) PACU patients with anticipated overnight stay.: In this study investigators will recruit patients that meet the following criteria:
  * Inclusion Criteria:
    * ≥18 years old undergoing non-cardiac surgery
    * Post-operative patients admitted to the PACU and expected to stay in the hospital for at least overnight
    * Receiving supplemental oxygen via face mask in the PACU
    * On continuous SpO2 saturation monitoring
    * Receiving standard postoperative of care
  * Exclusion Criteria:
    * Requirement for any form of postoperative invasive ventilatory support
    * Patients receiving only local or topical anesthesia
    * Day/outpatient surgery
    * Unable to cooperate with the application of the study device
    * Surgical/nursing/anesthesia staff suggest no study-related monitoring because of medical situation
  Interventions: Device: Linshom Continuous Predictive Respiratory Monitoring

INTERVENTIONS:
Device: Linshom Continuous Predictive Respiratory Monitoring — Observational study. Monitoring of Linshom, pulse oximetry and capnography data with comparison to current standard of care.
  Other Names: Pulse Oximetry, Capnography

SUMMARY:
Investigators will enroll 320 patients who will undergo non-cardiac surgery, receive supplemental oxygen via face mask, and will be on a continuous pulse oximetry monitor in the Post Anesthesia Care Unit (PACU). The enrollment criteria were adapted from a previous study that showed SpO2 values seriously underestimated the severity of post-operative hypoxemia in patients with and without specific risk factors for hypoxemia. Research personnel will screen and ensure that each subject meets the enrollment criteria, and the informed consent is properly executed. Upon arrival to the PACU, each subject will be fitted with oxygen mask containing the Linshom sensor, which will be connected to a Linshom monitor for data collection. A side stream capnography line will be connected to the same face mask and the capnography data will be collected on the Zoe Medical 740 SELECT™ monitor. Additionally, two pulse oximeters will be applied to the same hand (non- NIBP arm), one of which will be connected to a hospital monitor (SoC) and the other to a Zoe Medical 740 SELECT™ monitor. The Linshom and 740 SELECT™ monitors will collect data once every second.

Research personnel will then initiate the Linshom CPRM baseline mode and begin recording any clinical intervention (e.g., medications, oxygen delivery change, and stimulation upon detection of changes in patient's condition) that is performed by the PACU staff, paying close attention to, and recording of time at which those interventions occurred. Data collection will be performed throughout the subject's entire PACU stay. The CPRM data collection will be performed passively while the patient is monitored via SoC and will not interfere with clinical interventions that may take place during the data collection. Clinical staff in the PACU will be blinded to the Linshom CPRM data as well as pulse oximetry (non-SOC monitor) and capnography data collected.

DETAILED DESCRIPTION:
Linshom Medical (Linshom) has developed the FDA-cleared Continuous Predictive Respiratory Monitor (CPRM) a small and inexpensive sensor and monitor that provides continuous real-time tracking of these critical indicators of RDE. Linshom technology is based on our novel Linshom thermal sensor which is regulated by a thermoelectric cooler utilizing a proprietary control loop process. Respiration state is measured via temperature change throughout a patient's inspiratory/expiratory cycle. This delivers a respiratory signature allowing for continuous measurement of RR, relative Tidal Volume (rTV), relative Minute Ventilation (rMV), seconds since last breath (SSLB), and inspiratoryexpiratory (I/E) ratio. The CPRM solves existing unmet needs mentioned above with a small, portable, and inexpensive sensor and monitor that tracks RR, rTV, rMV (calculation of RR x rTV), seconds since last breath (SSLB), and I:E ratio in real time and continuously. These parameters are crucial in monitoring of patients suffering from both acute and chronic respiratory illness. Linshom offers an OR-quality respiratory profile at the patient bedside, which allows health care providers to promptly diagnose emerging respiratory decline and intervene with appropriate medical care.

In Phase I, investigators will conduct a clinical study in 145 post-operative patients comparing Linshom's CPRM to current SOC (clinical attention + pulse oximetry) and capnography. We will collect SOC, CPRM and capnography data simultaneously from each patient to demonstrate the ability of Linshom CPRM to identify Respiratory Depression Episodes in advance of SOC and/or capnography.

In Phase II, investigators will conduct a continuation of the phase I clinical study until the enrollment for this phase (175 patients) is reached, which would give an adequate statistical power for development of the Linshom CPRM alarm function.

Specific aims:

* Aim 1: Demonstrate that Linshom CPRM is able to identify RDE earlier than pulse oximetry and capnography.

  o Outcome: Investigators expect to successfully demonstrate that Linshom CPRM is capable of identifying RDE in advance of pulse oximetry and capnography by performing statistical analyses (non-inferiority and superiority hypothesis tests).
* Aim 2: Identify parameters and threshold values for the alarm function of Linshom CPRM for RR, rTV percent change, rMV percent change, I:E ratio and SSLB.

  * Outcome: Investigators will identify Linshom CPRM parameters and threshold values with high predictive abilities for RDE. These parameters and threshold values will be incorporated into future product to alert for clinicians and allow them to provide timely interventions to patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old undergoing non-cardiac surgery
* Post-operative patients admitted to the PACU and expected to stay in the hospital for at least overnight
* Receiving supplemental oxygen via face mask in the PACU
* On continuous SpO2 saturation monitoring
* Receiving standard postoperative of care

  • Exclusion Criteria:
* Requirement for any form of postoperative invasive ventilatory support
* Patients receiving only local or topical anesthesia
* Day/outpatient surgery
* Unable to cooperate with the application of the study device
* Surgical/nursing/anesthesia staff suggest no study-related monitoring because of medical situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted at The Ohio State University Wexner Medical Center (OSUWMC) where about 9% of the surgical procedures will go to the ICU or other non-PACU location and 20% will go home same day (within 24 hours). Based on previous trial data from OSUWMC, investigators expect gender to be ~50% male, 76% white and 23% non-white with an age distribution of 1/3 < 60 years of age and 2/3 > 60 years of age. This enrollment criteria makes the study results generalizable; population balanced and supports enrollment.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-09-28 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of Linshom CPRM to pulse oximetry with respect to the time (in minutes) prior to RDE that it was predicted that an RDE would occur. | 6-12 months
  The primary analysis will be to assess non-inferiority of Linshom to pulse oximetry with respect to the time (in minutes) prior to RDE that it was predicted that an RDE would occur.This analysis will be performed on patients with RDE. The statistical test to be used will be a paired t-test for non-inferiority of means.

SECONDARY OUTCOMES:
Superiority of Linshom CPRM to pulse oximetry, capnography and pulse oximetry + capnography with respect to the time (in minutes) prior to RDE that it was predicted that an RDE would occur. | Months 12-24
  Under the same assumptions of mean difference and standard deviation of the paired difference as for Phase I above, but with a -1 minute noninferiority margin, then a sample size of 128 subjects with RDE has 80% power to claim noninferiority of Linshom to pulse oximetry (i.e., 80% power to reject the above null hypothesis) at a one-sided 0.025 level of significance. Assuming prevalence of RDE in the PACU population is 40%, then 320 subjects will be enrolled in Phase I and II combined to achieve128 subjects with RDE for the Phase I + II combined primary analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Linshom Medical, Inc., Ellicott City, Maryland
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Data and specimens will only be shared with individuals who are members of the IRB approved research team or approved for sharing as described in this IRB protocol.

REFERENCES:
- [Result] Andersen LW, Berg KM, Chase M, Cocchi MN, Massaro J, Donnino MW; American Heart Association's Get With The Guidelines((R))-Resuscitation Investigators. Acute respiratory compromise on inpatient wards in the United States: Incidence, outcomes, and factors associated with in-hospital mortality. Resuscitation. 2016 Aug;105:123-9. doi: 10.1016/j.resuscitation.2016.05.014. Epub 2016 May 30. PMID 27255952
- [Result] Andersen LW, Kim WY, Chase M, Berg KM, Mortensen SJ, Moskowitz A, Novack V, Cocchi MN, Donnino MW; American Heart Association's Get With the Guidelines((R)) - Resuscitation Investigators. The prevalence and significance of abnormal vital signs prior to in-hospital cardiac arrest. Resuscitation. 2016 Jan;98:112-7. doi: 10.1016/j.resuscitation.2015.08.016. Epub 2015 Sep 9. PMID 26362486
- [Result] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Result] Overdyk FJ, Carter R, Maddox RR, Callura J, Herrin AE, Henriquez C. Continuous oximetry/capnometry monitoring reveals frequent desaturation and bradypnea during patient-controlled analgesia. Anesth Analg. 2007 Aug;105(2):412-8. doi: 10.1213/01.ane.0000269489.26048.63. PMID 17646499
- [Result] Taenzer AH, Pyke JB, McGrath SP, Blike GT. Impact of pulse oximetry surveillance on rescue events and intensive care unit transfers: a before-and-after concurrence study. Anesthesiology. 2010 Feb;112(2):282-7. doi: 10.1097/ALN.0b013e3181ca7a9b. PMID 20098128
- [Result] Wadhwa V, Gonzalez AJ, Selema K, Feldman R, Lopez R, Vargo JJ. Novel device for monitoring respiratory rate during endoscopy-A thermodynamic sensor. World J Gastrointest Pharmacol Ther. 2019 Jul 18;10(3):57-66. doi: 10.4292/wjgpt.v10.i3.57. PMID 31598389
- [Result] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Result] Khanna AK, Sessler DI, Sun Z, Naylor AJ, You J, Hesler BD, Kurz A, Devereaux PJ, Saager L. Using the STOP-BANG questionnaire to predict hypoxaemia in patients recovering from noncardiac surgery: a prospective cohort analysis. Br J Anaesth. 2016 May;116(5):632-40. doi: 10.1093/bja/aew029. PMID 27106966
- [Result] May AM, Kazakov J, Strohl KP. Predictors of Intraprocedural Respiratory Bronchoscopy Complications. J Bronchology Interv Pulmonol. 2020 Apr;27(2):135-141. doi: 10.1097/LBR.0000000000000619. PMID 31478940
- [Result] Fu ES, Downs JB, Schweiger JW, Miguel RV, Smith RA. Supplemental oxygen impairs detection of hypoventilation by pulse oximetry. Chest. 2004 Nov;126(5):1552-8. doi: 10.1378/chest.126.5.1552. PMID 15539726
- [Result] Niesters M, Mahajan RP, Aarts L, Dahan A. High-inspired oxygen concentration further impairs opioid-induced respiratory depression. Br J Anaesth. 2013 May;110(5):837-41. doi: 10.1093/bja/aes494. Epub 2013 Jan 4. PMID 23293275